CLINICAL TRIAL: NCT06746168
Title: Infiltration of Local Anesthetics Between the Popliteal Artery and Capsule of the Knee (iPACK) With Femoral Triangle Block (TFB) Versus Surgical Local Infiltration Analgesia (LIA) in Unilateral Total Knee Arthroplasty (TKA): A Multicenter Double-blind, Prospective Randomized Controlled Study.
Brief Title: BLOCK-study: Better Local Orthopedic Pain Control After Knee Arthroplasty
Acronym: BLOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, MD, PhD, Jessa Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/178
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Knee Arthroplasty, Total
Keywords: iPACK; Femoral Triangle Block; Local infiltration analgesia; knee arthoplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iPACK with Femoral Triangle Block (FTB) (Active Comparator): Patients undergoing an unillateral total kneearthroplasty will receive the anesthetic combination iPACK with FTB.
  Interventions: Procedure: Locoregional anesthesia
- Surgical Local Infiltration Analgesia (LIA) (Active Comparator): Patients undergoing an unillateral total kneearthroplasty will receive the surgical LIA.
  Interventions: Procedure: Local Anesthetic Ropivacaine

INTERVENTIONS:
Procedure: Locoregional anesthesia — The FTB + iPACK group will receive 12 ml 0,5% ropivacaine for the FTB and 20 ml of ropivacaine 0.5% for the iPACK block under US guidance after spinal anesthesia
  Arms: iPACK with Femoral Triangle Block (FTB)
Procedure: Local Anesthetic Ropivacaine — The control group (LIA) will receive 120 ml 0.25% ropivacaine for surgical LIA placement.
  Arms: Surgical Local Infiltration Analgesia (LIA)

SUMMARY:
The goal of this study is to compare the anesthetic combination iPACK with femoral triangle block versus surgical LIA for unilateral TKA. We hypothesize that an iPACK block with femoral triangle block is non-inferior to surgical LIA. Furthermore, due to visualization of the relevant neural and vascular structures, the risk of accidental popliteal block, nerve damage or LAST with (a blindly performed) LIA could theoretically be reduced.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* BMI 17-35 kg/m2
* Patient is able to give informed consent
* Patient is scheduled for TKA

Exclusion Criteria:

* Refusal of patient
* Inability to communicate due to language or neurologic barriers
* Bilateral TKA or unilateral knee arthroplasty
* Chronic opioid use (including partial opioid agonists) + chronic pain patients:
* Use of atypical analgesics (gabapentin, pregabalin, …)
* History of Sudeck atrophy
* History of >3 chronic pain consultations
* Contraindications for spinal anesthesia
* Patient refusal
* Local infection
* Aberrant coagulation (according to the latest ESRA guidelines)
* Severe spinal canal stenosis
* Intracranial hypertension
* History of neurological injury in the affected limb
* Contraindications for local anesthetics
* Allergy for local anesthetics
* Absolute contraindications for NSAIDs or paracetamol
* Proven allergy for NSAID's (including ASA syndrome) or paracetamol
* Severe renal function impairment (eGFR <30 ml/min/1.73 m2)
* Active or recent (<6 months) history of gastric ulcera/perforations/bleeding
* Crohn disease or colitis ulcerosa
* Liver function impairment or severe renal function impairment (eGFR <30 ml/min/1.73 m2)
* Pregnancy or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain score at mobilization at 8 hour postoperatively | 8 hours postoperatively
  The NRS pain score will be determined immediately after mobilizing patients from the bed to their seat at 8 hour postoperatively

SECONDARY OUTCOMES:
NRS pain at movement for the first 24 hours | 24 hours postoperatively
  The Area Under the Curve for the NRS pain scores at movement will be evaluated at 4h-6h-8h-12h-24h after the surgery
NRS pain at rest for the first 24 hours | 24 hours postoperatively
  The Area Under the Curve for the NRS pain scores at rest will be evaluated at 4h-6h-8h-12h-24h after the surgery
Rate of popliteal block 8 hours after surgery | 8 hours postoperatively
  the incidence of a popliteal block will be assessed 8 hours after surgery
Functional recovery: timed up and go test | Baseline, 24 hours and 48 hours after surgery
  Patients have to sit in a standard sitting chair, stand up from the chair, walk 3 meters, get back to the chair and sit down. A cut-off of 13.5 seconds or longer indicates higher risk of falls, normal values depend on age.
Functional recovery: 30-second sit-to-stand-chair test | Baseline, 24 hours and 48 hours after surgery
  In the 30 seconds sit-to-stand chair test, patients must try to stand up and sit down again from a chair as much as possible in the 30 seconds time interval. Arms need to be crossed and may not be used to stand up. Normal values vary according to age.
Quality of Life: Short-form 36 (SF-36) questionnaire | Baseline, 3 months, 6 months
  The SF-36 questionaire is the most widely used health-related quality of life score. They identified 8 health concepts to be scored in the SF-36: Physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal/emotional problems, general mental health, social functioning, energy/fatigue/vitality and general health perceptions.
Quality of Life: WOMAC questionnaire | Baseline, 3 months, 6 months
  The WOMAC-index (Western Ontario and McMaster Universities Osteoartritis index) evaluates the broader functional impact of (initially) osteoarthritis but is now often used as quality of life indicator after total knee arthroplasty.
Incidence of rescue blocks | 8 to 12 hours after the spinal anesthesia
  In case of persistent pain (NRS > 6) despite the abovementioned regimen (cut-off: need for more than 20 opioid oral morphine milligrams equivalents over 12h), a rescue femoral triangle (10-15 ml ropivacaine 0.5%) and iPACK block (20 ml ropivacaine 0.5%) can be applied 8-12h after the initial locoregional procedure.
Need for rescue analgesia | during hospital stay, an average of 3 days
  The need and dose for rescue analgesia (oral morphine equivalents) will be calculated
Time to be fit for discharge | during hospital stay, an average of 3 days
  - Time to be fit for discharge as defined by:
  * Oral pain medication only
  * Independent walking (with crutches)
  * Full oral diet
  * Hemodynamically and respiratory (no need for oxygen) stable
  * No drains or urinary catheters This will be assess until day of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium